CLINICAL TRIAL: NCT02765867
Title: A Single-Dose, Open-Label Study of Depot Buprenorphine (RBP-6000) in Opioid-Dependent Individuals
Brief Title: Single-dose, Study of RBP-6000 in Opioid Dependent Individuals
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Indivior Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RB-US-10-0011
Record Dates: First submitted 2016-05-04; First posted 2016-05-09 (Estimated); Last update posted 2016-05-09 (Estimated); Status verified 2016-05

CONDITIONS: Opioid Use Disorder
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- RBP-6000 (Experimental): A single dose of RBP-6000 will be administered on Study Day 1
  Interventions: Drug: RBP-6000

INTERVENTIONS:
Drug: RBP-6000 — A single injection of RBP-6000 containing a low dose of buprenorphine in the Atrigel delivery system

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability and pharmacokinetic profile of an injection of RBP-6000.

DETAILED DESCRIPTION:
This is an open-label, single-center, first-in-human study, designed to evaluate the safety, tolerability and pharmacokinetic (PK) profile of a single subcutaneous (SC) injection of RBP-6000 in opioid dependent subjects. Enrollment will begin with 6 subjects, and additional subjects will not be enrolled until safety through Day 4 has been reviewed and analyzed. Subjects will remain in a residential unit through Day 30 post-injection and will continue with visits to the clinical unit until Day 85 or plasma buprenorphine levels are below 100 pg/mL, whichever comes later. The expected maximum duration of participation for each subject (including screening) is 120 days.

Safety will be assessed by adverse events, electrocardiograms, clinical laboratory assessments, local injection site tolerability and vital signs. PK will be assessed by measuring concentrations of buprenorphine and norbuprenorphine in plasma. The need for rescue medication will be assessed using clinical judgment along with information provided by the COWS scores.

ELIGIBILITY:
Inclusion Criteria:

* If female, must be surgically sterile or two-years post-menopausal and have a negative pregnancy test. Subjects should take reasonable precautions during the study to avoid pregnancy by agreeing to remain abstinent or to practice double-barrier forms of birth control from study screening through the last dose of study medication.
* Meet Diagnostic and Statistical Manual of Mental Disorders, 4th Edition, Text Revision (DSM-IV-TR) criteria for opioid dependence and who are seeking opioid-dependence treatment with methadone.
* Willing to cooperate with study procedures and provide written informed consent prior to start of any study procedures.
* Agree not to take any buprenorphine product (other than RBP-6000) throughout their participation in the study.
* Body mass index of ≥ 18 to ≤ 33 kg/m2.
* Total bilirubin < 2.5 mg/dL (51 μmol/L), alanine aminotransferase (ALT) or aspartate aminotransferase (AST) < 3 × the upper limit of normal (ULN), serum creatinine < 2 x ULN, or international normalized ratio (INR) ≤ 2.0.
* Normal or no clinically significant ECG findings at screening

Exclusion Criteria:

* Require ongoing opioid therapy for pain or other chronic medical conditions.
* Additionally, individuals who answer "yes" to both of the following questions will be excluded from participation: A) Throughout our lives, most of us have had pain from time to time (such as minor headaches, sprains, and toothaches). Have you had pain other than those kinds of pain today? B) If yes, has the pain persisted for three months or more?
* Currently dependent by DSM-IV-TR criteria on any substance other than opioids, caffeine, or nicotine.
* Positive urine screen at intake for barbiturates, benzodiazepines, buprenorphine, or methadone.
* History or presence of clinically significant cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, oncologic, or psychiatric disease or any other condition that, in the opinion of the study physician, would jeopardize the safety of the subject.
* Clinically significant abnormal finding on physical exam or in medical history; serology positive for HIV, hepatitis B or C [HBV antigen S positive, acute HBsAg and IgM antiHBc Chronic HCV antibody HCV, HCV RNA- acute: HCV RNA (PCR)].
* History or presence of allergic or adverse response (including rash or anaphylaxis) to buprenorphine, methadone, or the ATRIGEL Delivery System.
* Donation of more than 250 mL of blood or plasma, or participation in another clinical trial, within 30 days prior to signing of the informed consent document for this study.
* Currently (during past 30 days from the signing of the informed consent document) engaged in opioid agonist, partial agonist, or antagonist treatment, or require on-going prescription or over-the-counter medications that are clinically relevant P450 3A4 inducers or inhibitors [azole antifungals (e.g. ketoconazole), macrolide antibiotics (e.g. erythromycin),].
* Reporting taking buprenorphine within 30 days of screening.
* Significant traumatic injury, major surgery or open biopsy within the prior 4 weeks.
* Subjects who have been previously excluded from participation or previously enrolled into the study.
* Subjects who are unable, in the opinion of the Principal Investigator and/or the medically responsible physician, to comply fully with the study requirements.
* Subjects who have participated in another investigational product trial within 30 days of screening.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2010-11; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
To assess the incidence of treatment emergent adverse events (safety and tolerability) of a single SC injection of RBP-6000 in subjects with opioid dependence. | Day 1 to Day 85
  The frequency of all adverse events (AE) and serious adverse events (SAE) deemed to be related to treatment.

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) for buprenorphine and norbuprenorphine | Day 1 through Day 85
  PK samples to be collected to determine Cmax over the post-injection period
Time to occurrence of Cmax (Tmax) for buprenorphine and norbuprenorphine | Day 1 through Day 85
  PK samples to be collected to determine Tmax over the post-injection period
Area under the plasma concentration versus time curve (AUC) for buprenorphine and norbuprenorphine | Day 1 through Day 85
  AUC to be measured from time 0 to the last sampling time post-injection at which concentrations were at or above the limit of quantitation

CONTACTS AND LOCATIONS:
Locations (1):
- Scientific Clinical Research, Fort Lauderdale, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided